CLINICAL TRIAL: NCT01824186
Title: A Randomized Controlled Trial Comparing Post-operative Pain in Single-incision Laparoscopic Cholecystectomy Versus Conventional Laparoscopic Cholecystectomy
Brief Title: Trial Comparing Pain in Single-incision Laparoscopic Cholecystectomy Versus Conventional Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NHG DSRB 2009/00434
Record Dates: First submitted 2013-03-21; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Cholelithiasis; Choledocholithiasis; Cholecystolithiasis; Pancreatitis; Cholangitis
MeSH Terms: conditions — Cholelithiasis; Choledocholithiasis; Cholecystolithiasis; Pancreatitis; Cholangitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SILC (Experimental): Subjects in this arm were randomized to undergo single-incision laparoscopic cholecystectomy, through a transumbilical incision
  Interventions: Procedure: SILC
- LC (Active Comparator): Subjects in this arm were randomized to undergo conventional 4-port laparoscopic cholecystectomy. Wound sites at umbilicus, right hypocondrium, epigastrium and right flank
  Interventions: Procedure: LC

INTERVENTIONS:
Procedure: SILC — Underwent single-incision laparoscopic cholecystectomy
  Other Names: Single-incision laparoscopic cholecystectomy
  Arms: SILC
Procedure: LC — Underwent conventional 4-port laparoscopic cholecystectomy
  Other Names: Conventional laparoscopic cholecystectomy
  Arms: LC

SUMMARY:
This study aims to evaluate post-operative pain in single-incision laparoscopic cholecystectomy (SILC) versus the conventional four port technique (LC). The investigators hypothesize that SILC is non-inferior in post-operative pain.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* presence of symptomatic gallstones
* American Society of Anesthesiologists (ASA) score 1 or 2
* informed consent

Exclusion Criteria:

* active acute cholecystitis
* previous open upper abdominal surgery
* bleeding disorders

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Post-operative pain 4 hours | 4 hours post-operative
  To evaluate post-operative pain in single-incision laparoscopic cholecystectomy vs the conventional 4 port technique. Measured at both umbilical and extra-umbilical sites, at rest and on movement. Visual analogue scale, from 1-10.
Post-operative pain 24 hours | 24 hours post-operative
  To evaluate post-operative pain in single-incision laparoscopic cholecystectomy vs the conventional 4 port technique. Measured at both umbilical and extra-umbilical sites, at rest and on movement. Visual analogue scale, from 1-10.
Post-operative pain 14 days | 14 days post-operative
  To evaluate post-operative pain in single-incision laparoscopic cholecystectomy vs the conventional 4 port technique. Measured at both umbilical and extra-umbilical sites, at rest and on movement. Visual analogue scale, from 1-10.
Post-operative pain 6 months | 6 months post-operative
  To evaluate post-operative pain in single-incision laparoscopic cholecystectomy vs the conventional 4 port technique. Measured at both umbilical and extra-umbilical sites, at rest and on movement. Visual analogue scale, from 1-10.

SECONDARY OUTCOMES:
Procedural complications | 6 months
  To evaluate complications between single-incision laparoscopic cholecystectomy vs the conventional four port technique. Conducted via telephone interview and review of hospital records in the intervening period
Operative duration | following skin closure
  To evaluate operative duration between single-incision laparoscopic cholecystectomy vs the conventional four port technique
Subject satisfaction | 14 days and 6 months
  To evaluate subject satisfaction between single-incision laparoscopic cholecystectomy vs the conventional four port technique. Measured on a Likert scale, from 1-5 (1 least satisfied, 5 most satisfied)
Return to function | 14 days
  To evaluate post-operative return to function following surgery, between single-incision laparoscopic cholecystectomy vs the conventional four port technique. Measured as days taken to independent toileting, and independently obtaining meals as a surrogate measure of function

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kin Yong Chang, FRCS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Chang SK, Wang YL, Shen L, Iyer SG, Madhavan K. A randomized controlled trial comparing post-operative pain in single-incision laparoscopic cholecystectomy versus conventional laparoscopic cholecystectomy. World J Surg. 2015 Apr;39(4):897-904. doi: 10.1007/s00268-014-2903-6. PMID 25446490